CLINICAL TRIAL: NCT06058611
Title: Effects of a Personalised and Tailored Computerised Cognitive Stimulation Programme Versus Stimulating Leisure Activities in Older Adults with Mild Cognitive Impairment and Subjective Cognitive Impairment: Randomised Controlled Trial
Brief Title: Effects of a Computerised Cognitive Stimulation Versus Stimulating Leisure Activities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Isabel Gómez-Soria, Assistant professor doctor, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U
Record Dates: First submitted 2023-09-16; First posted 2023-09-28 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment; Randomized Controlled Trial; Subjective Cognitive Impairment
Keywords: Mild Cognitive Impairment; Older adults; Elderly; Randomized Controlled Trial; Cognitive Stimulation; Cognitive Intervention; Cognitively Stimulating Leisure Activities; Leisure Activities; Subjective Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Parallel allocation Two intervention group (GI1 and GI2) and a control group (CG) with the same characteristics are included
Who Masked: Outcomes Assessor
Masking Description: The professionals responsible for the assessments will be blinded and will be different from the professionals carrying out the intervention. Both will be trained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group 1 (GI1) (Experimental): Intervention group 1 (IG1) will carry out personalised and adapted computerised cognitive stimulation (CE) through the stimulus platform; 30 minutes/day, 5 days/week, 8 weeks; 40 sessions. The following will be worked on: memory, orientation, language, praxis, gnosis, calculation, perception, logical reasoning, attention-concentration and executive functions.
  Interventions: Other: Cognitive stimulation
- Intervention group 2 (GI2) (Experimental): Intervention group 2 (IG2) will perform between 2 and 5 cognitively stimulating leisure activities for 8 weeks. These leisure activities will be selected from the adapted version of the Karp et al. 2006 questionnaire (Karp et al., 2006) taking into account the three components of leisure activities (mental, physical and social). The questionnaire contains 29 activities.
  In addition to indicating which cognitively stimulating leisure activities they perform on a weekly basis, participants in IG2 will indicate their daily frequency (< 30 min, 30min-1 hour, 1-2 hours, > 2 hours), commenting on whether they have carried them out individually or in a group. It will also be taken into account whether these activities were previously carried out according to their stage of life.
  Interventions: Other: Stimulating leisure activities
- Control Group (CG) (No Intervention): The control group (CG) will not receive any intervention during the study period.

INTERVENTIONS:
Other: Cognitive stimulation — Cognitive stimulation through the stimulus platform; 30 minutes/day, 5 days/week, 8 weeks; 40 sessions. The following will be worked on: memory, orientation, language, praxis, gnosis, calculation, perception, logical reasoning, attention-concentration and executive functions.
  Arms: Intervention group 1 (GI1)
Other: Stimulating leisure activities — Intervention group 2 (IG2) will perform between 2 and 5 cognitively stimulating leisure activities for 8 weeks. These leisure activities will be selected from the adapted version of the Karp et al. 2006 questionnaire (Karp et al., 2006) taking into account the three components of leisure activities (mental, physical and social). The questionnaire contains 29 activities.
  In addition to indicating which cognitively stimulating leisure activities they perform on a weekly basis, participants in IG2 will indicate their daily frequency (< 30 min, 30min-1 hour, 1-2 hours, > 2 hours), commenting on whether they have carried them out individually or in a group. It will also be taken into account whether these activities were previously carried out according to their stage of life.
  Arms: Intervention group 2 (GI2)

SUMMARY:
The aim of the study is to evaluate, at the level of global cognition, cognitive neuroconstructs, memory, verbal fluency, ADLs, IADLs, symptoms of depression and anxiety, the effectiveness of a personalised and adapted computerised cognitive stimulation programme (GI1) implemented from Primary Care versus stimulating leisure activities (GI2), in older adults aged 50 years and over with mild cognitive impairment and subjective cognitive impairment living in the community.

DETAILED DESCRIPTION:
A randomised controlled trial (RCT) will be conducted. The sample will consist of 59 participants aged 50 years and older, all of whom are patients in primary care practices.

Intervention Intervention group 1 (IG1) will carry out personalised and adapted computerised CE through the stimulus platform; 30 minutes/day, 5 days/week, 8 weeks; 40 sessions. The following will be worked on: memory, orientation, language, praxis, gnosis, calculation, perception, logical reasoning, attention-concentration and executive functions. Stimulus is a CE platform, which allows individualised intervention through the use of ICTs with different populations.

Intervention group 2 (IG2) will perform between 2 and 5 cognitively stimulating leisure activities for 8 weeks. These leisure activities will be selected from the adapted version of the Karp et al. 2006 questionnaire (Karp et al., 2006) taking into account the three components of leisure activities (mental, physical and social). The questionnaire contains 29 activities [1) reading, 2) arts and crafts, 3) crosswords and word search puzzles, 4) interest in politics, 5) playing cards or chess, 6) visiting the second home, 7) attending courses, 8) watching television, 9) going to the theatre or concerts, 10) playing sports, 11) going to exhibitions or museums, 12) meeting friends, 13) walking, 14) listening to the radio, 15) travelling, 16) gardening, 17) painting, drawing or taking photos, 18) participating in family or charity activities, 19) outdoor activities, 20) collecting stamps or other items, 21) cooking, 22) writing, 23) doing housework, 24) attending religious activities, 25) playing musical instruments, 26) playing solitaire, 27) following the stock market or investing, 28) playing bingo, 29) singing].

In addition to indicating which cognitively stimulating leisure activities they perform on a weekly basis, participants in IG2 will indicate their daily frequency (< 30 min, 30min-1 hour, 1-2 hours, > 2 hours), commenting on whether they have carried them out individually or in a group. It will also be taken into account whether these activities were previously carried out according to their stage of life.

The control group (CG) will not receive any intervention during the study period. At the end of the study, the control group will be offered to participate in either of the following two interventions.

There will be a pre-intervention, post-intervention assessment and two follow-ups at 6 and 12 months. Firstly, an assessment protocol will be used with ad hoc socio-demographic variables, referring to clinical characteristics and in relation to lifestyle. These variables will be collected in a socio-health record. In addition, if participants do not have a diagnosis of MCI, the MEC-35 will be used to apply the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years old, resident in the community.
* Diagnosis of MCI or having between 24 and 27 points on the MEC-35 (this score seems to indicate the presence of MCI) (Calero, M. D and Navarro, 2006).
* Subjective cognitive impairment (score between 28-31 points on the MEC-35) (Gómez-Soria et al. 2023)

Exclusion Criteria:

* Institutionalisation.
* Taking acetylcholinesterase inhibitors as they may act on global cognition and/or cognitive functions.
* Sensory deficits (deafness and blindness) preventing intervention.
* Agitation.
* Having received cognitive stimulation in the last 12 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Lobo Cognitive Mini-Test (MEC-35) | Post-intervention (1 week), 3 months, 6 months, 12 months
  The MEC-35 is one of the most widely used short cognitive tests for the study of cognitive abilities in the primary care setting. The MEC-35 assesses eight cognitive functions: temporal and spatial orientation (10 items), fixation memory (3 items), attention (3 items), calculation (5 items), short-term memory (3 items) and language and praxis (11 items) (Lobo et al. 1999) (figure 1). Its sensitivity is 89.8% and its specificity 83.9% (Calero MD, Navarro E, Robles P, 2000). Unlike the MMSE, the MEC-35 includes a series of three digits to repeat two similar items in reverse order. Subtraction is performed 3 by 3 from 30, instead of 7 by 7 from 100 (Folstein et al., 1975).

SECONDARY OUTCOMES:
Test of Memory Alteration (T@M) | Post-intervention (1 week), 3 months, 6 months, 12 months
  The maximum score for the T@M is 50 points; one point is awarded for each correct answer. All questions are oral and have only one possible answer. There are 5 sub-tests: encoding (5 points), orientation (10 points), semantic (15 points), free recall (10 points) and guided recall (10 points). It assesses temporal orientation and memory (episodic, textual and semantic). A score of 36 points has a sensitivity of 0.93 and a specificity of 1 (Rami et al., 2009). Its results are slightly influenced by educational level, so the cut-off points are 36/37 and 37/38 for subjects with <8 years and ≥8 years of education, respectively (Carnero-Pardo et al., 2011).

OTHER OUTCOMES:
Set-Test (S-T) | Post-intervention (1 week), 3 months, 6 months, 12 months
  The Set-Test (S-T) assesses semantic fluency across four categories: colours, animals, fruits and cities. Scores range from 0 to 40, with 0 being the minimum score and 40 the maximum. The cut-off point is 27 points, and a lower score indicates dementia. This questionnaire has a sensitivity of 79% and a specificity of 82% (Pascual Millán, LF, Martínez Quiñones, JV, Modrego Pardo, P, Mostacero Miguel, E, López del Val, J, Morales Asín, 1990).
Activities of Daily Living Questionnaire T-ADLQ | Post-intervention (1 week), 3 months, 6 months, 12 months
  The Activities of Daily Living Questionnaire T-ADLQ assesses 7 ADL areas: self-care (6 items), home care and management (6 items), work and leisure (4 items), shopping and money (3 items), travel (3), communication (5 items) and technology (5 items) (Figure 4). Each item has a score, where 0 is no problem for the activity up to 3 indicating that the activity cannot be performed. It is flexible in that it does not score aspects that are not part of the patient's activities (Muñoz-Neira et al., 2012). The internal consistency of the 33 items is high (Cronbach's α coefficient 0.848). The internal consistency of each of the 7 subscales was either low (Cronbach's α value of 0.396 for Travel and 0.539 for Employment and Leisure) or high (Cronbach's α value of 0.688 for Shopping and Money and 0.739 for Employment and Leisure ,780 for Home Care, 0.739 for Self-Care Activities and 0.862 for the Technology subscale) (Terwee et al., 2007).
Lawton and Brody scale (L-B) | Post-intervention (1 week), 3 months, 6 months, 12 months
  Autonomy in eight IADLs required for independent living will be assessed with the Lawton and Brody (L-B) scale. Scores range from 0 (dependent) to 8 (independent). The sensitivity of the scale is 57% and its specificity 82% when a respondent observes dependence in three activities (Pfeffer et al., 1982).
15-item version of the Yesavage Geriatric Depression Scale (GDS-15) | Post-intervention (1 week), 3 months, 6 months, 12 months
  The 15-item version of the Yesavage Geriatric Depression Scale (GDS-15) will be used to assess symptoms of depression. This scale is considered suitable for community-dwelling older adults. Scores range from 0 to 15, and a total score > 5 is interpreted as "probable depression". In older adults, with a cut-off point of 5 points, the sensitivity is 71.8% and the specificity 78.2% (Marc et al., 2008).
Goldberg anxiety subscale | Post-intervention (1 week), 3 months, 6 months, 12 months
  To assess the level of anxiety, the Goldberg anxiety subscale with nine dichotomous response items (yes/no answers) will be administered. A separate score is given for each scale, with one point per affirmative response. The cut-off value is ≥ 4 for the anxiety subscale, indicating "probable anxiety". This scale shows a specificity of 91% and a sensitivity of 86% (Goldberg et al., 1988).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud Arrabal, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lobo A, Saz P, Marcos G, Dia JL, de la Camara C, Ventura T, Morales Asin F, Fernando Pascual L, Montanes JA, Aznar S. [Revalidation and standardization of the cognition mini-exam (first Spanish version of the Mini-Mental Status Examination) in the general geriatric population]. Med Clin (Barc). 1999 Jun 5;112(20):767-74. Spanish. PMID 10422057
- [Background] Calero MD, Navarro E, Robles P, Garcia-Berben TM. [[Validity of the Cognitive Mini-Exam of Lobo et al. for the detection of dementia-associated cognitive deterioration] ]. Neurologia. 2000 Oct;15(8):337-42. Spanish. PMID 11143500
- [Background] Rami L, Bosch B, Valls-Pedret C, Caprile C, Sanchez-Valle Diaz R, Molinuevo JL. [Discriminatory validity and association of the mini-mental test (MMSE) and the memory alteration test (M@T) with a neuropsychological battery in patients with amnestic mild cognitive impairment and Alzheimer's disease]. Rev Neurol. 2009 Aug 16-31;49(4):169-74. Spanish. PMID 19621317
- [Background] Carnero-Pardo C, Espejo-Martinez B, Lopez-Alcalde S, Espinosa-Garcia M, Saez-Zea C, Hernandez-Torres E, Navarro-Espigares JL, Vilchez-Carrillo R. Diagnostic accuracy, effectiveness and cost for cognitive impairment and dementia screening of three short cognitive tests applicable to illiterates. PLoS One. 2011;6(11):e27069. doi: 10.1371/journal.pone.0027069. Epub 2011 Nov 2. PMID 22073256
- [Background] Pascual Millan LF, Martinez Quinones JV, Modrego Pardo P, Mostacero Miguel E, Lopez del Val J, Morales Asin F. [The set-test for diagnosis of dementia]. Neurologia. 1990 Mar;5(3):82-5. Spanish. PMID 2361045
- [Background] Munoz-Neira C, Lopez OL, Riveros R, Nunez-Huasaf J, Flores P, Slachevsky A. The technology - activities of daily living questionnaire: a version with a technology-related subscale. Dement Geriatr Cogn Disord. 2012;33(6):361-71. doi: 10.1159/000338606. Epub 2012 Jul 11. PMID 22797087
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Pfeffer RI, Kurosaki TT, Harrah CH Jr, Chance JM, Filos S. Measurement of functional activities in older adults in the community. J Gerontol. 1982 May;37(3):323-9. doi: 10.1093/geronj/37.3.323. PMID 7069156
- [Background] Marc LG, Raue PJ, Bruce ML. Screening performance of the 15-item geriatric depression scale in a diverse elderly home care population. Am J Geriatr Psychiatry. 2008 Nov;16(11):914-21. doi: 10.1097/JGP.0b013e318186bd67. PMID 18978252
- [Background] Goldberg D, Bridges K, Duncan-Jones P, Grayson D. Detecting anxiety and depression in general medical settings. BMJ. 1988 Oct 8;297(6653):897-9. doi: 10.1136/bmj.297.6653.897. PMID 3140969
- [Background] Karp A, Paillard-Borg S, Wang HX, Silverstein M, Winblad B, Fratiglioni L. Mental, physical and social components in leisure activities equally contribute to decrease dementia risk. Dement Geriatr Cogn Disord. 2006;21(2):65-73. doi: 10.1159/000089919. Epub 2005 Nov 23. PMID 16319455